CLINICAL TRIAL: NCT05620875
Title: The Association Between Delivered Oxygen and Cerebral Impact During the Use of Cardiopulmonary Bypass.
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06630-01
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cardiac; Arteriosclerosis; Aortic Valve Disease
MeSH Terms: conditions — Arteriosclerosis; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples Without DNA — Cerebral injury markers in blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group with DO2i <280 ml/min/m2 during cardiopulmonary bypass
  Interventions: Diagnostic Test: Cerebral injury markers; Diagnostic Test: Cerebral oximetry index
- Group with DO2i >280 ml/min/m2 during cardiopulmonary bypass
  Interventions: Diagnostic Test: Cerebral injury markers; Diagnostic Test: Cerebral oximetry index

INTERVENTIONS:
Diagnostic Test: Cerebral injury markers — Blood tests at given time points perioperatively.
Diagnostic Test: Cerebral oximetry index — Cerebral oximetry index measurements with the aid of Near Infrared Spectroscopy

SUMMARY:
Investigating the connection between delivered oxygen index and cerebral impact with COx (cerebral oximetry index) och cerebral injury markers during the routine use of cardiopulmonary bypass.

DETAILED DESCRIPTION:
The research subjects are to be treated with CPB with according to local standards (perfusion index 2.4 x body surface area). While measuring impact on cerebral autoregulation with the aid of Near InfraRed Spectroscopy (NIRS) and brain injury markers in blood, research subjects depending on initial hemoglobin value, will divide into two subgroups: one with DO2I of >280 ml/min/m2, and one with DO2I of <280 ml/min/m2.

DO2I will during CPB be calculated using the patient data monitoring system Metavision.

With a correlation analysis between NIRS and MAP (mean arterial pressure) a COx (Cerebral Oxymetry Index) r-value can indicate impact on cerebral autoregulation with values >0.3 - 0.5 during use of CPB 4.

Brain injury markers (Tau, Glial Fibrillary Acidic Protein (GFAP), Neurospecific Enolase (NSE)) are collected during 5 occasions during the first 24 hours and then once per day for 4 days, as well as markers for AKI (S-Creatinine) in some extent.

Registrations during the intensive care regarding delirium, stroke or other neurological impact will also be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for CABG and/or AVR

Exclusion Criteria:

* Former diagnosed neurological insults, carotid stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 120 research subjects scheduled for coronary arterial bypass grafting surgery and/or aortic valve replacement in Uppsala University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
COx | 24 hours
  COx (Cerebral Oximetry Index; correlation between rSO2 values (INVOS) and mean artery pressure) that indicated impact on cerebral autoregulation on DO2 index values below set limits of 280 ml/m2/min.
Brain injury markers; tau, GFAP, NSE | 96 hours
  Brain injury markers that indicate cerebral neuronal damage on DO2 index values below set limits of 280 ml/m2/min.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Henrik Grinnemo, Adj. Prof., Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden